CLINICAL TRIAL: NCT03631667
Title: Ultralow Dose PAH Binary Mixture Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oregon State University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH); Lawrence Livermore National Laboratory (Other); Pacific Northwest National Laboratory (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Williams, Professor, Oregon State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LPI-8554; R01ES028600 (NIH)
Record Dates: First submitted 2018-08-08; First posted 2018-08-15 (Actual); Results first posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Environmental Exposure
Keywords: Benzo[a]pyrene; Accelerator Mass Spectrometry; Polycyclic Aromatic Hydrocarbons; Phenanthrene
MeSH Terms: interventions — phenanthrene

STUDY DESIGN:
Masking Description: Deidentified samples will be analyzed by AMS at Lawrence Livermore National Laboratory and the pharmacokinetics determine at Pacific Northwest National Laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 50 ng dose and 50 ng dose plus 1250 ng phenanthrene (Experimental): Cycle 1: Capsule containing 50 ng (5.4 nCi) [14C]-benzo[a]pyrene (BaP).
  Cycle 2: Capsule containing 50 ng (5.4 nCi) [14C]-benzo[a]pyrene (BaP) and 1250 phenanthrene.
  At least 3 weeks will pass between cycles as a washout period.
  Interventions: Drug: [14C]-benzo[a]pyrene; Drug: [14C]-benzo[a]pyrene plus phenanthrene

INTERVENTIONS:
Drug: [14C]-benzo[a]pyrene — Oral micro-dose (50 ng) (5.4 nCi)
  Other Names: Carcinogenic PAH environmental pollutant
Drug: [14C]-benzo[a]pyrene plus phenanthrene — Oral micro-dose of 50 ng (5.4 nCi) [14C]-benzo[a]pyrene plus 1250 ng phenanthrene
  Other Names: Binary mixture of carcinogenic PAH and non-carcinogenic PAH

SUMMARY:
Evaluation of the pharmacokinetics for [14C]-benzo[a]pyrene ([14C]-BaP) and metabolites in plasma and urine over 48 hours following a 50 ng dose (5.4 nCi) alone or with 1250 ng phenanthrene.

DETAILED DESCRIPTION:
The pharmacokinetics for [14C]-BaP and metabolites will be assessed by UHLPC-Accelerator Mass Spectrometry (AMS, Lawrence Livermore National Laboratory) in plasma and urine collected over 48 hours following oral doses of 50 ng dose (5.4 nCi) alone or with 1250 ng phenanthrene. Metabolite profiles and kinetics of elimination are predicted to be consistent with a BaP physiologically based pharmacokinetic (PBPK) model developed by Pacific Northwest National Laboratory (PNNL). A non-smoker, not exposed occupationally, receives 270-700 ng of BaP daily; about 95% dietary. The WHO has set an estimated safe daily lifetime (70 year/70 Kg individual, cancer endpoint) exposure to BaP of 42-350 ng. This protocol represents de minimus risk.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-65 (inclusive)
* If female, must be post-menopausal or have had surgical sterilization to eliminate any possibility for fetal exposure
* Willing to defer blood donation for one month before, throughout, and one month after completion of study activities
* Willing to avoid consuming cruciferous vegetables, I3C or DIM supplements, smoked or cured meat or cheeses, or charcoal-grilled meats for 2 weeks prior to and during each study cycle (gas grilled foods acceptable)

Exclusion Criteria:

* Smoker (tobacco or other substances) or use of smokeless tobacco in past 3 months or living with smoker
* Regular use of medications that affect gut motility or nutrient absorption (e.g. cholestyramine, sucralfate, orlistat, pro- or anti-motility agents)
* History of gastrointestinal surgery (e.g. bariatric surgery, cholecystectomy) or gastrointestinal disorder (Crohn's disease, celiac disease, IBS, or colitis)
* Current or history of kidney or liver disease
* Prior high-dose 14C exposure from medical tests. (micro-dose 14C exposure not exclusionary)
* Occupational PAH exposure (e.g. roofers, asphalt pavers, fire-fighters, etc.)
* Regular use of indole-3-carbinol or DIM dietary supplements

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon State University, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified samples sent to Lawrence Livermore National Laboratory Deidentified data sent to Pacific Northwest National Laboratory

RESULTS

PARTICIPANT FLOW:
Groups:
- 50 ng Dose and 50 ng Dose Plus 1250 ng Phenanthrene: Capsule containing 50 ng (5.4 nCi) [14C]-benzo[a]pyrene (BaP). Capsule containing 50 ng (5.4 nCi) [14C]-benzo[a]pyrene (BaP) and 1250 phenanthrene. At least 3 weeks must pass between each capsule dose administration.
  [14C]-benzo[a]pyrene: Oral micro-dose (50 ng) (5.4 nCi)
  [14C]-benzo[a]pyrene plus phenanthrene: Oral micro-dose of 50 ng (5.4 nCi) [14C]-benzo[a]pyrene plus 1250 ng phenanthrene
Period: Overall Study
Arm/Group | 50 ng Dose and 50 ng Dose Plus 1250 ng Phenanthrene
Started | 8 (8 participants consented to participate. 3 participants voluntarily withdrew prior to beginning the study protocol (no BaP doses administered).)
Completed | 5
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | 50 ng Dose and 50 ng Dose Plus 1250 ng Phenanthrene
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration of 14C-BaP Cmax
Description: Determination of highest concentration of 14C-BaP in plasma. Blood samples collected at 0 (baseline), 0.25, 0.5, 1, 2, 3, 4, 8, 24, and 48 hour after dosing. All time points were used to determine Cmax.
Time Frame: 0-48 hours for each of 2 dosing cycles, with a washout period of 3 weeks between the dosing cycles
Measure: Mean (Standard Deviation); unit: fg [14C]-BaP/mL plasma
Groups:
- 50 ng Dose and 50 ng Dose Plus 1250 ng Phenanthrene: Cycle 1: Capsule containing 50 ng (5.4 nCi) [14C]-benzo[a]pyrene (BaP).
  Cycle 2: Capsule containing 50 ng (5.4 nCi) [14C]-benzo[a]pyrene (BaP) and 1250 phenanthrene.
  At least 3 weeks will pass between cycles as a washout period.
  [14C]-benzo[a]pyrene: Oral micro-dose (50 ng) (5.4 nCi)
  [14C]-benzo[a]pyrene plus phenanthrene: Oral micro-dose of 50 ng (5.4 nCi) [14C]-benzo[a]pyrene plus 1250 ng phenanthrene
Arm/Group | 50 ng Dose and 50 ng Dose Plus 1250 ng Phenanthrene
Number analyzed (Participants) | 5
fg [14C]-BaP/mL plasma
  50 ng [14C]-BaP | 7.07 (4.89)
  50 ng [14C]-BaP plus 1250 ng phenanthrene | 1.60 (0.86)

2. Primary Outcome: Time at Highest Plasma Concentration of 14C-BaP Tmax
Description: Determination of time at which plasma concentration of 14C-BaP is highest. Blood samples collected at 0 (baseline), 0.25, 0.5, 1, 2, 3, 4, 8, 24, and 48 hour after dosing. All time points were used to determine Tmax.
Time Frame: 0-48 hours for each of 2 dosing cycles, with a washout period of 3 weeks between the dosing cycles
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | 50 ng Dose and 50 ng Dose Plus 1250 ng Phenanthrene
Number analyzed (Participants) | 5
hour
  50 ng [14C]-BaP | 1.1 (1.1)
  50 ng [14C]-BaP plus 1250 ng phenanthrene | 1.7 (1.3)

3. Secondary Outcome: Area Under Plasma Concentration of 14C-BaP Versus Time Curve AUC
Description: Integration of concentration of 14C-BaP in plasma over time. Blood samples collected at 0 (baseline), 0.25, 0.5, 1, 2, 3, 4, 8, 24, and 48 hour after dosing. All time points were used to determine AUC.
Time Frame: 0-48 hours for each of 2 dosing cycles, with a washout period of 3 weeks between the dosing cycles
Measure: Mean (Standard Deviation); unit: fg [14C]-BaP/mL plasma x hour
Arm/Group | 50 ng Dose and 50 ng Dose Plus 1250 ng Phenanthrene
Number analyzed (Participants) | 5
fg [14C]-BaP/mL plasma x hour
  50 ng [14C]-BaP | 17.88 (9.56)
  50 ng [14C]-BaP plus 1250 ng phenanthrene | 10.07 (9.32)

4. Secondary Outcome: Rate of Elimination of 14C-BaP (Half Life)
Description: Determination of constants for rate of elimination of 14C-BaP from plasma. Blood samples collected at 0 (baseline), 0.25, 0.5, 1, 2, 3, 4, 8, 24, and 48 hour after dosing. All time points were used to determine half-life.
Time Frame: 0-48 hours for each of 2 dosing cycles, with a washout period of 3 weeks between the dosing cycles
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | 50 ng Dose and 50 ng Dose Plus 1250 ng Phenanthrene
Number analyzed (Participants) | 5
hour
  50 ng [14C]-BaP | 4.78 (4.45)
  50 ng [14C]-BaP plus 1250 ng phenanthrene | 3.92 (4.12)

ADVERSE EVENTS:
Time Frame: 48.5 hours for each of 2 dosing cycles with a 3-week washout period between the dosing cycles. Participants were assessed for adverse events 15 minutes prior to the [14c]-BaP dose administration (time= 0 hour) until 15 minutes after the final blood sample collection time point (time = 48 hour) and removal of the peripheral IV catheter.
Description: The definitions of adverse event and serious adverse event used to determine incidence are consistent with clinicaltrials.gov definitions. Each participant was verbally asked about the occurrence of adverse events at each clinical visit by the research nurse.
Arm/Group | 50 ng Dose and 50 ng Dose Plus 1250 ng Phenanthrene
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT03631667/Prot_SAP_ICF_000.pdf